CLINICAL TRIAL: NCT05553574
Title: Inhibitory Capabilities Among Women With Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Shir Berebbi, PhD Student, Hebrew University of Jerusalem
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SB1
Record Dates: First submitted 2021-05-26; First posted 2022-09-23 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Food Response; Food Stop; Food Response-inhibition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Food response (Experimental)
  Interventions: Behavioral: Stop signal food task
- Food stop (Experimental)
  Interventions: Behavioral: Stop signal food task
- Food response-inhibition (Experimental)
  Interventions: Behavioral: Stop signal food task

INTERVENTIONS:
Behavioral: Stop signal food task — The participants need to classify pictures of food and not food. They were asked to hold their response if they see a white frame around the picture.

SUMMARY:
The goal of the study is to increase the flexible behavior toward food via inhibition training among restrained eaters. The expectation is that the train will increase food consumption, decrease food-related anxiety and affect implicit attitudes towards palatable foods

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of restrained eaters
* Adults ages 18-40

Exclusion Criteria:

* Current history or diagnosis of the following according to the criteria of the DSM-5:

Schizophrenia, schizoaffective disorder, hallucinations, unspecified psychotic disorder (NOS), a mental disorder due to acquired head injury, bipolar disorder, mental disorder as a result of organic development.

* Abuse or addiction to drugs and alcohol.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Main outcome | one hour
  The participants will increase food consumption,decrease food-related anxiety and affect implicit attitudes towards palatable foods

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew university of Jerusalem, Jerusalem, Israel